CLINICAL TRIAL: NCT01328925
Title: Double-blind, Placebo-controlled Study of Nitazoxanide Suspension in the Treatment of Rotavirus Disease in Children
Brief Title: Efficacy Study of Nitazoxanide Suspension in the Treatment of Rotavirus Disease in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Romark Laboratories L.C. (Industry)
Responsible Party: Celine Rossignol, MS, Romark Laboratories, L.C.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RM02-3022
Record Dates: First submitted 2011-03-29; First posted 2011-04-05 (Estimated); Last update posted 2011-04-05 (Estimated); Status verified 2011-04

CONDITIONS: Rotavirus Infection; Viral Gastroenteritis Due to Rotavirus
Keywords: Rotavirus; Viral gastroenteritis; Gastroenteritis
MeSH Terms: conditions — Rotavirus Infections; Gastroenteritis | interventions — nitazoxanide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nitazoxanide Oral Suspension (Experimental): Nitazoxanide Oral Suspension 100 mg/5 ml
  Interventions: Drug: Nitazoxanide
- Placebo Oral Suspension (Placebo Comparator): Placebo Oral Suspension
  Interventions: Drug: Nitazoxanide

INTERVENTIONS:
Drug: Nitazoxanide — Nitazoxanide Oral Suspension dose based on age:
  Age <12 months- 7.5 mg/kg by mouth twice daily for 3 days; Age 12-47 months- 100 mg/5 ml by mouth twice daily for 3 days; Age 48-72 months- 200 mg/10 ml by mouth twice daily for 3 days
  Other Names: Alinia; NTZ

SUMMARY:
The purpose of this study is to determine the effectiveness of nitazoxanide suspension compared to placebo in treating rotavirus disease in pediatric patients less than 6 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Age < 6 years.
* Patients with diarrhea (defined as 3 or more liquid stools per day).
* Stool positive for rotavirus by ELISA.

Exclusion Criteria:

* Other identified causes of diarrhea at screening (pathogenic protozoa, bacteria, viruses or lactose intolerance).
* Serious systemic disorders incompatible with the study.

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2005-12; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Time from first dose to resolution of symptoms. | Up to 14 days
  Resolution of all gastrointestinal symptoms associated with viral diarrhea at enrollment including abdominal pain or tenderness, distention, etc. with the patient not requiring anti-motility or other palliative treatment. Symptom resolution must be maintained for at least 48 hours to be considered valid.

SECONDARY OUTCOMES:
Time from first dose to virologic response | Up to 14 days
  Daily stool samples will be analyzed by ELISA for the presence of rotavirus. Virologic response is defined by a negative ELISA stool test for rotavirus on 2 consecutive days.
Time from first dose to hospital discharge | Up to 14 days
  For hospitalized patients, the study will monitor the time in hours from the first dose of study medication to discharge from the hospital.
Volume of oral rehydration solutions consumed | Up to 14 days
Frequency of intravenous rehydration required | Up to 14 days
Stool weight | Up to 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Mona Abu-Zekry, MD, Principal Investigator — Cairo University Children's Hospital
Locations (1):
- Cairo University Children's Hospital, Cairo, Egypt